CLINICAL TRIAL: NCT07125651
Title: Prevalence of Gastrointestinal Bleeding in Ischemic Heart Disease Patients Undergoing Single Compared to Dual Antiplatelet Treatment
Brief Title: Gastrointestinal Bleeding is Blood Loss in the Digestive Tract, Classified as Upper or Lower. Ischemic Heart Disease is Due to Blocked Heart Arteries. Antiplatelet Drugs Help Prevent Heart Attacks But Increase GI Bleeding Risk, Especially When Used Together as Dual Therapy.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Antar Mohamed, Dr, Assiut University
Other Study IDs: GIB in IHD patients on APT
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gastro Intestinal Bleeding; Ischaemic Heart Diseases; Antiplatelet Drugs; Antiplatelet Drug-related Gastrointestinal Injury
Keywords: Gastrointestinal bleeding; GIB; ischemic heart disease; IHD; Antiplatelet therapy; SAPT; DAPT
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal bleeding is blood loss in the digestive tract, classified as upper or lower. Ischemic heart disease is due to blocked heart arteries. Antiplatelet drugs help prevent heart attacks but increase GI bleeding risk, especially when used together as dual therapy. This study aims to compare the prevalence and risk of gastrointestinal bleeding in ischemic heart disease patients on single versus dual antiplatelet therapy, and to explore strategies for reducing gastrointestinal bleeding in these patients, enhancing treatment safety without compromising cardiovascular protection.

DETAILED DESCRIPTION:
Gastrointestinal (GI) bleeding refers to blood loss within the gastrointestinal tract, including the esophagus, stomach, small and large intestines, rectum, and anus. It is classified as upper GI bleeding-originating proximal to the ligament of Treitz (esophagus, stomach, first and second parts of the duodenum)-and lower GI bleeding, which originates distal to this ligament (remaining duodenum, jejunum, ileum, colon, rectum, and anus). GI bleeding may be acute, with sudden and severe blood loss, or chronic, involving slow, recurrent bleeding that is less obvious but still clinically significant.

Ischemic heart disease (IHD) is caused by reduced blood flow to the heart muscle due to narrowing or blockage of the coronary arteries, mainly from atherosclerosis. This can result in chest pain, heart attacks, and other cardiovascular complications.

Antiplatelet drugs, such as aspirin and clopidogrel, inhibit platelet aggregation to prevent blood clots and are essential in IHD management. Single antiplatelet therapy (SAPT) uses one agent, while dual antiplatelet therapy (DAPT) combines two agents for stronger protection against thrombotic events.

Both SAPT and DAPT improve cardiovascular outcomes in IHD patients, with SAPT commonly used for long-term prevention and DAPT recommended after acute coronary events or interventions.

Antiplatelet drugs, like aspirin and clopidogrel, increase GI bleeding risk by inhibiting platelet aggregation, impairing clot formation, and, in the case of aspirin, directly irritating the stomach lining, making it easier for ulcers or erosions to bleed. The risk is higher with dual therapy.

This study aims to compare the prevalence and risk of gastrointestinal bleeding in ischemic heart disease patients on single versus dual antiplatelet therapy, and to explore strategies for reducing gastrointestinal bleeding in these patients, enhancing treatment safety without compromising cardiovascular protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients (aged 18 years old and older) who were diagnosed ischemic heart disease on single or dual antiplatelet therapy and developed gastrointestinal bleeding (manifestation of hematemesis, melena or bleeding per rectum).

Exclusion Criteria:

* Patients on anticoagulant.
* Patients with bleeding tendencies.
* Individuals with other comorbidities.
* patients with acute coronary syndrome.
* Uncooperative patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (aged 18 years old and older) who were diagnosed ischemic heart disease on single or dual antiplatelet therapy and developed gastrointestinal bleeding (manifestation of hematemesis, melena or bleeding per rectum).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gastrointestinal bleeding in ischemic heart disease patients undergoing single compared to dual antiplatelet treatment | Baseline
  Gastrointestinal bleeding is blood loss in the digestive tract, classified as upper or lower. Ischemic heart disease is due to blocked heart arteries. Antiplatelet drugs help prevent heart attacks but increase GI bleeding risk, especially when used together as dual therapy.

REFERENCES:
- [Background] Abraham NS, Hlatky MA, Antman EM, Bhatt DL, Bjorkman DJ, Clark CB, Furberg CD, Johnson DA, Kahi CJ, Laine L, Mahaffey KW, Quigley EM, Scheiman J, Sperling LS, Tomaselli GF; ACCF/ACG/AHA. ACCF/ACG/AHA 2010 Expert Consensus Document on the concomitant use of proton pump inhibitors and thienopyridines: a focused update of the ACCF/ACG/AHA 2008 expert consensus document on reducing the gastrointestinal risks of antiplatelet therapy and NSAID use: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. Circulation. 2010 Dec 14;122(24):2619-33. doi: 10.1161/CIR.0b013e318202f701. Epub 2010 Nov 8. No abstract available. PMID 21060077
- [Background] Lanas A, Wu P, Medin J, Mills EJ. Low doses of acetylsalicylic acid increase risk of gastrointestinal bleeding in a meta-analysis. Clin Gastroenterol Hepatol. 2011 Sep;9(9):762-768.e6. doi: 10.1016/j.cgh.2011.05.020. Epub 2011 Jun 6. PMID 21699808
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2016 Sep 6;68(10):1082-115. doi: 10.1016/j.jacc.2016.03.513. Epub 2016 Mar 29. No abstract available. PMID 27036918
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Lanas A, Garcia-Rodriguez LA, Polo-Tomas M, Ponce M, Alonso-Abreu I, Perez-Aisa MA, Perez-Gisbert J, Bujanda L, Castro M, Munoz M, Rodrigo L, Calvet X, Del-Pino D, Garcia S. Time trends and impact of upper and lower gastrointestinal bleeding and perforation in clinical practice. Am J Gastroenterol. 2009 Jul;104(7):1633-41. doi: 10.1038/ajg.2009.164. Epub 2009 May 5. PMID 19574968
- [Background] Libby P, Theroux P. Pathophysiology of coronary artery disease. Circulation. 2005 Jun 28;111(25):3481-8. doi: 10.1161/CIRCULATIONAHA.105.537878. PMID 15983262
- [Background] Longstreth GF. Epidemiology and outcome of patients hospitalized with acute lower gastrointestinal hemorrhage: a population-based study. Am J Gastroenterol. 1997 Mar;92(3):419-24. PMID 9068461